CLINICAL TRIAL: NCT01693822
Title: A-PREDICT: A Phase II Study Of Axitinib In Metastatic Renal Cell Cancer in Patients Unsuitable for Nephrectomy
Brief Title: A Phase II Study of Axitinib in Patients With Metastatic Renal Cell Cancer Unsuitable for Nephrectomy
Acronym: A-PREDICT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Pfizer (Industry); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2011/10033
Record Dates: First submitted 2012-08-06; First posted 2012-09-26 (Estimated); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Clear-cell Metastatic Renal Cell Carcinoma
Keywords: metastatic renal cell carcinoma; predominant clear cell histology; Unsuitable for nephrectomy; unsuitable for 'watch and wait' policy
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib (Experimental): Axitinib - oral tablet twice daily until disease progression. Starting dose 5mg.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Axitinib treatment Axitinib is an oral VEGF-receptor inhibitor. Patients are prescribed a starting dose of 5mg twice daily, escalating to 10mg in absence of dose limiting toxicities.
  Patients should stop axitinib treatment one week prior to day 1 week 9 percutaneous research biopsy of the primary renal tumour and restart 2-3 days post biopsy.
  Doses should be taken approximately 12 hours apart and patients should be instructed to take their doses at approximately the same times each day.
  Dose adjustments, including dose increase or dose reduction, are permitted and should be based on clinical judgement and the guidelines provided in the protocol.
  Other Names: AG-013736

SUMMARY:
A-PREDICT is a study of axitinib in patients with metastatic renal cell carcinoma unsuitable for nephrectomy (as judged by the treating clinician) to evaluate efficacy, safety, toxicity and changes in biomarkers during therapy. Axitinib will given twice daily by mouth according to tolerability of treatment, for as long as patients are deriving clinical benefit. Blood and tumour tissue samples will be taken prior to and during therapy to evaluate biomarkers of treatment response. The primary clinical objective of this study is to define the activity of axitinib given to patients with metastatic renal cell carcinoma unsuitable for nephrectomy.

DETAILED DESCRIPTION:
A-PREDICT is a single arm, single agent, open label, multicentre, phase II study of axitinib in patients with metastatic renal cell carcinoma of predominant clear cell histology and unsuitable for debulking nephrectomy (as judged by the treating clinician). Patients who have provided consent and have satisfied the eligibility criteria will be registered into the trial.

The starting dose of axitinib will be 5 mg twice daily by mouth, escalating to a maximum of 10mg twice daily by mouth according to tolerability of treatment, for as long as patients are deriving clinical benefit. Treatment will be paused for one week prior to percutaneous biopsy of the primary on day 1 week 9. Disease progression will be evaluated according to RECIST v1.1 criteria 8 weeks after commencing treatment, at 8 weekly intervals to 6 months and 3 monthly thereafter. Blood and tumour tissue samples will be taken prior to and during therapy to evaluate biomarkers of treatment response. Nephrectomy will be carried out on any patient who becomes suitable in the opinion of the treating clinician during the course of the trial. Where possible, tissue samples will be taken from resected specimens. Response to axitinib in marker lesions will be correlated with changes in biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic renal cell carcinoma of predominant clear cell histology
2. Unsuitable for nephrectomy
3. Unsuitable for 'watch and wait' policy
4. No prior systemic therapy for renal cell carcinoma
5. Measurable metastatic disease using RECIST v1.1
6. Life expectancy 12 weeks or greater
7. ECOG performance status 0 or 1
8. Adequate organ function as defined by serum aspartate transaminase (AST) or serum alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to liver metastases; total serum bilirubin ≤1.5 x ULN
9. Adequate haematological function as defined by absolute neutrophil count (ANC) ≥1500/μL, platelets ≥75,000/μL, haemoglobin ≥9.0 g/dL and prothrombin time (PT) ≤1.5 x ULN
10. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥ 60 mL/min;
11. Urinary protein <2+ by urine dipstick.
12. No evidence of pre-existing uncontrolled hypertension
13. Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.
14. Willingness and ability to comply with study procedures, including tumour biopsies.
15. Written informed consent

Exclusion Criteria:

1. The presence of intracranial disease, unless stable >6 months. In the case of a solitary brain metastasis which has been resected, there must be evidence of a disease-free interval of at least 3 months post-surgery. All patients previously treated for brain metastases must be stable off corticosteroid therapy for at least 28 days.
2. The presence of active second malignancy.
3. Women who are pregnant or are breastfeeding. Female patients must be surgically sterile, be postmenopausal, or must agree to use effective contraception during the period of therapy.
4. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy.
5. Current signs or symptoms of severe progressive or uncontrolled hepatic, endocrine, pulmonary disease other than directly related to RCC.
6. Gastrointestinal abnormalities including:

   1. inability to take oral medication;
   2. requirement for intravenous alimentation;
   3. prior surgical procedures affecting absorption including total gastric resection;
   4. treatment for active peptic ulcer disease in the past 6 months;
   5. active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
   6. malabsorption syndromes.
7. Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (see section 8.12, concomitant therapy).
8. Current use or anticipated need for treatment with drugs that are known CYP3A4 or CYP1A2 inducers (see section 8.12, concomitant therapy).
9. Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access device or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
10. Active seizure disorder, spinal cord compression, or carcinomatous meningitis.
11. Any of the following within 12 months prior to study entry: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
12. Deep vein thrombosis or pulmonary embolism within 6 months prior to study entry.
13. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
14. Known galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-10; Primary Completion 2017-03 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Larkin, Principal Investigator — Royal Marsden Hospital London
Locations (11):
- United Kingdom (11):
  - Royal Surrey County Hospital, Guildford, Surrey
  - Royal Marsden Hospital - Sutton, London, Sutton
  - Addenbrooke's Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Free Hospital, London
  - Guy's Hospital, London
  - Royal Marsden Hospital, London
  - Christie Hospital, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, together with a data dictionary defining each field in the set, will be made available to other researchers on request, subject to the approval of a formal data access request in accordance with the ICR-CTSU data and sample access policy. Trial documentation including the protocol are available on request by contacting apredict-icrctsu@icr.ac.uk Formal requests for data sharing are considered in line with ICR-CTSU procedures. Requests are via a standard proforma describing the nature of the proposed research and extent of data requirements. Contact apredict-icrctsu@icr.ac.uk or visit the link below for further information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available to researchers following the formal review and approval of a data access request in accordance with the ICR-CTSU data and sample access policy.
Access Criteria: Completion and approval of a data access request form as stated above.
URL: https://www.icr.ac.uk/our-research/centres-and-collaborations/centres-at-the-icr/clinical-trials-and-statistics-unit/working-with-us/data-sharing

REFERENCES:
- See also: ICR-CTSU trial page — https://www.icr.ac.uk/our-research/centres-and-collaborations/centres-at-the-icr/clinical-trials-and-statistics-unit/our-research/clinical-trials/a-predict

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: Axitinib - oral tablet twice daily until disease progression. Starting dose 5mg.
  Axitinib: Axitinib treatment Axitinib is an oral VEGF-receptor inhibitor. Patients are prescribed a starting dose of 5mg twice daily, escalating to 10mg in absence of dose limiting toxicities.
  Patients should stop axitinib treatment one week prior to day 1 week 9 percutaneous research biopsy of the primary renal tumour and restart 2-3 days post biopsy.
  Doses should be taken approximately 12 hours apart and patients should be instructed to take their doses at approximately the same times each day.
  Dose adjustments, including dose increase or dose reduction, are permitted and should be based on clinical judgement and the guidelines provided in the protocol.
Period: Overall Study
Arm/Group | Axitinib
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: ITT
Arm/Group | Axitinib
Number analyzed (Participants) | 65
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.5 [56.7 to 69.0]
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 8
  50-59 years | 19
  60-69 years | 26
  70+ years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Histological type [Count of Participants; unit: Participants]
  Clear cell | 62
  Clear cell and chromophobe | 2
  Clear cell and sarcomatoid component | 1
Fuhrman grade [Count of Participants; unit: Participants]
  G1 - inconspicuous nucleoli at ×400 magnification and basophilic (low-grade) | 2
  G2 - clearly visible nucleoli at ×400 magnification and eosinophilic (low-grade) | 26
  G3 - clearly visible nucleoli at ×100 magnification (high grade) | 21
  G4 - extreme pleomorphism or rhabdoid and/or sarcomatoid morphology (high grade and most aggressive) | 2
  Unobtainable | 14
Motzer Score [Count of Participants; unit: Participants] — Risk factors for Motzer score evaluation include :
  Time from diagnosis to systemic treatment <1 year Measured ~1 month after stopping anticoagulation Hemoglobin < Lower Limit of Normal Calcium >10mg/dL (>2.5 mmol/L) LDH > 1.5x Upper Limit of Normal Performance status <80% (Karnofsky)
  Participants
    Intermediate risk (1-2 risk factors) | 50
    High risk (3+ risk factors) | 15

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Progression at 6 Months
Description: The proportion of study participants alive and progression free at 6 months (day 1 week 25 visit). Progression will be measured from the date of study entry (registration date) until the first date of either death or confirmed progressive disease according to RECIST v1.1 (https://recist.eortc.org/recist-1-1-2/). Patients alive and free from progression will be censored at the date of last follow-up. The proportion of patients progression free at 6 months will be reported with 95% confidence interval. In addition, progression free survival will be presented using the Kaplan Meier product limit method with median progression free survival reported. A blinded central review of CT scans will be conducted for verification purposes.
Time Frame: 6 months
Population: Reporting group
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Axitinib
Number analyzed (Participants) | 65
Percentage | 58.5 [45.6 to 70.6]

2. Secondary Outcome: Best Overall Response
Description: Best overall response (one of Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD) throughout the treatment period according to RECIST v1.1 (https://recist.eortc.org/recist-1-1-2/).
Time Frame: From registration, during treatment and up to 30 days after treatment discontinuation. Patients remain on treatment until disease progression assessed up to 106 months.
Population: Reporting group
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 65
Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 19
  Stable Disease (SD) | 29
  Progressive Disease (PD) | 16

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) will be measured from the date of registration until first date of either death or confirmed progressive disease according to RECIST 1.1. Time to last follow-up will be used if patient has not progressed or died and PFS time for the patient will be considered censored. A Kaplan Meier graph and median survival time will be presented.
Time Frame: From the date of registration until first date of either death or confirmed progressive disease from any cause, whichever came first, assessed up to 106 months.
Population: Reporting group
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib
Number analyzed (Participants) | 65
Months | 63.1 [50.2 to 74.7]

4. Secondary Outcome: Overall Survival
Description: Overall survival will be measured from the date of registration until the date of death due to any cause. Time to last follow-up will be used if patient has not died and survival time for the patient will be considered censored.
Time Frame: From the date of registration until the date of death due to any cause, up to 106 months.
Population: Reporting group
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Axitinib
Number analyzed (Participants) | 65
Months | 19.7 [9.2 to 37.2]

5. Secondary Outcome: Safety and Toxicity of Axitinib (by NCI CTC Grading Version 4)
Description: Progression of the malignancy was not reported as a serious adverse event. Hospitalisation due to signs and symptoms of malignancy progression was not reported as a serious adverse event. Occurrences are counted as any subject reporting a particular AE at a visit where toxicity was assessed.
Time Frame: Treatment duration (at least 4 weekly, and again at disease progression), up to 106 months.
Population: This population contains all patients who received at least one dose of axitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 64
Participants
  Total subjects affected by serious adverse events subjects affected / exposed | 26
  number of deaths (all causes) | 62
  number of deaths resulting from adverse events | 3

6. Secondary Outcome: Number of Patients Who Become Suitable for Nephrectomy as a Consequence of Therapy With Axitinib
Description: The proportion of patients who undergo nephrectomy following registration as a result of treatment with axitinib will be reported with 95% confidence intervals.
Time Frame: Study duration (assessed by clinician over treatment duration), up to 106 months.
Population: Reporting group
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 65
Participants | 9

ADVERSE EVENTS:
Time Frame: AEs were assessed up to 28 days after the patient discontinued study drug, up to 106 months.. All-Cause Mortality was assessed up to 106 months. Both were assessed from the date of registration.
Description: Progression of the malignancy was not reported as a serious adverse event. Hospitalisation due to signs and symptoms of malignancy progression was not reported as a serious adverse event. Occurrences are counted as any subject reporting a particular AE at a visit where toxicity was assessed.
Arm/Group | Axitinib
All-Cause Mortality (participants affected / at risk) | 62/64
Serious Adverse Events (participants affected / at risk) | 26/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (N=64)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Blood calcium increased (Psychiatric disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Hypophagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urosepsis (Renal and urinary disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (N=64)
Hot flush (Vascular disorders) | 4 (19)
Hypertension (Vascular disorders) | 60 (881)
Chest pain (General disorders) | 11 (15)
Fatigue (General disorders) | 61 (651)
Mucosal inflammation (General disorders) | 32 (157)
Oedema peripheral (General disorders) | 4 (9)
Pain (General disorders) | 11 (50)
Pyrexia (General disorders) | 10 (13)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (105)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 26 (190)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (145)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (22)
Insomnia (Psychiatric disorders) | 17 (99)
Mood altered (Psychiatric disorders) | 6 (9)
Alanine aminotransferase increased (Investigations) | 4 (8)
Blood alkaline phosphatase increased (Investigations) | 10 (22)
Blood creatinine decreased (Investigations) | 4 (11)
Blood creatinine increased (Investigations) | 8 (23)
Blood lactate dehydrogenase increased (Investigations) | 7 (25)
Blood magnesium decreased (Investigations) | 4 (13)
Gamma-glutamyltransferase increased (Investigations) | 8 (26)
Lymphocyte count decreased (Investigations) | 11 (49)
Platelet count increased (Investigations) | 6 (8)
Prothrombin time prolonged (Investigations) | 4 (9)
Weight decreased (Investigations) | 28 (166)
Wound complication (Injury, poisoning and procedural complications) | 4 (4)
Dizziness (Nervous system disorders) | 12 (44)
Dysgeusia (Nervous system disorders) | 28 (167)
Headache (Nervous system disorders) | 16 (35)
Neuralgia (Nervous system disorders) | 5 (7)
Neuropathy peripheral (Nervous system disorders) | 5 (8)
Paraesthesia (Nervous system disorders) | 6 (28)
Anaemia (Blood and lymphatic system disorders) | 13 (24)
Abdominal pain (Gastrointestinal disorders) | 26 (131)
Constipation (Gastrointestinal disorders) | 27 (189)
Diarrhoea (Gastrointestinal disorders) | 38 (434)
Dry mouth (Gastrointestinal disorders) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 15 (56)
Mouth ulceration (Gastrointestinal disorders) | 4 (14)
Nausea (Gastrointestinal disorders) | 38 (181)
Oral pain (Gastrointestinal disorders) | 6 (25)
Stomatitis (Gastrointestinal disorders) | 22 (90)
Vomiting (Gastrointestinal disorders) | 24 (79)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (54)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (31)
Palmar-plantar Erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 23 (217)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (10)
Rash (Skin and subcutaneous tissue disorders) | 20 (85)
Proteinuria (Renal and urinary disorders) | 38 (234)
Renal pain (Renal and urinary disorders) | 5 (11)
Hyperthyroidism (Endocrine disorders) | 4 (4)
Hypothyroidism (Endocrine disorders) | 28 (194)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (204)
Back pain (Musculoskeletal and connective tissue disorders) | 37 (236)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (16)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 20 (56)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 (16)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (71)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (33)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 (101)
Lower respiratory tract infection (Infections and infestations) | 7 (13)
Nasopharyngitis (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (10)
Decreased appetite (Metabolism and nutrition disorders) | 45 (243)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (41)
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 (34)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between principal investigators and the Sponsor (or its agents) that restricts the PIs rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT01693822/Prot_SAP_000.pdf